CLINICAL TRIAL: NCT00474201
Title: The Influence of Lopinavir/Ritonavir on Gemfibrozil Pharmacokinetics in Healthy Volunteers
Brief Title: Drug Interaction Study of Lopinavir/Ritonavir and Gemfibrozil
Acronym: GEM-PK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Principal Investigator, Scott Penzak, Pharm.D., Director, Clinical Pharmacokinetics research Laboratory, National Institutes of Health Clinical Center (CC)
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 070149; 07-CC-0149 CL006000-01 CC (Other: Clinical Center Z number)
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetic; HIV; Drug-Drug Interaction; Lopinavir/Ritonavir; Gemfibrozil; Healthy Volunteer; HV
MeSH Terms: interventions — Lopinavir; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemfibrozil PK without LPV/r (Sham Comparator): Subjects received a single 600 mg dose of gemfibrozil without concurrent lopinavir-ritonavir 400mg/100mg; this is the "control" arm of a crossover study design.
  Interventions: Drug: Gemfibrozil
- Gemfibrozil PK after 2 weeks of LPV/r (Experimental): Single dose (600 mg) Gemfibrozil pharmacokinetics (i.e. plasma concentrations collected over time to calculate area under the concentration vs. time curve) assessed after 14.5 days of lopinavir/ritonavir (400/100 mg twice daily) administration.
  Interventions: Drug: Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Lopinavir/Ritonavir — lopinavir 400 mg + ritonavir 100 mg twice daily for 2 weeks
  Other Names: lopinavir/ritonavir = Kaletra(TM)
  Arms: Gemfibrozil PK after 2 weeks of LPV/r
Drug: Gemfibrozil — Control arm (no intervention used in this arm)
  Other Names: gemfibrozil (Teva Pharmaceuticals)
  Arms: Gemfibrozil PK without LPV/r

SUMMARY:
This study will determine whether the protease inhibitor lopinavir/ ritonavir (Kaletra (Trademark)), which is used to treat HIV disease, lowers blood levels of the lipid-regulating drug gemfibrozil (Lopid (Trademark)) in HIV-negative healthy volunteers. Many patients with HIV infection who take protease inhibitors have abnormally high lipids (cholesterol and triglycerides). Gemfibrozil, commonly used to treat high triglycerides, often is not effective in HIV-infected patients taking protease inhibitors, possibly because of an interaction between the two medicines that causes a lowering of gemfibrozil's levels in the blood. Results from this study will give researchers information on whether lopinavir/ ritonavir affects the blood levels of gemfibrozil.

Healthy, normal volunteers between 18 and 65 years old who test negative for HIV may be eligible for this study.

On study day 1, subjects have a blood sample drawn from a catheter inserted into a vein in the arm to determine pre-dosing blood levels of gemfibrozil. They then take a gemfibrozil tablet and are given breakfast 30 minutes after taking the drug. Blood samples are obtained through the catheter at 0, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours after dosing to determine gemfibrozil levels at those intervals. At the end of 12 hours, the catheter is removed and the subject is discharged from the clinic. The next morning subjects return to the clinic for another blood sample, collected through a vein in the arm.

Subjects begin taking lopinavir/ ritonavir between 7 and 35 days after their first dose, depending on their schedule and the clinic schedule. On the fourteenth day of dosing subjects come to the clinic and are given a single dose of gemfibrozil, as on study day 1, and have breakfast 30 minutes later. Blood samples are collected to determine gemfibrozil levels just like on study days 1 and 2. An additional sample is collected for routine lab tests.

DETAILED DESCRIPTION:
Hyperlipidemia continues to be a common problem in individuals with HIV, particularly those receiving HIV protease inhibitors (PIs) or the nucleoside reverse transcriptase inhibitor, stavudine. PI-treated patients have been noted to have increases in low-density lipoprotein (LDL), triglycerides (TG), and total cholesterol compared to PI-treatment naive individuals. The prevalence of lipid abnormalities in patients receiving PI-containing therapy has been estimated at 27-57 percent; moreover, cardiovascular complications have begun to be revealed. Triglyceride elevations, in particular, are not only an independent risk factor for the development of coronary artery disease, but may also lead to pancreatitis. Despite treatment with fibric acid derivatives, such as gemfibrozil, TGs typically remain elevated above the upper limit of normal in HIV-infected subjects. One possible reason for persistently elevated TGs in these patients is reduced efficacy of their fibric acid therapy, which may result from an unrecognized drug-drug interaction. Fibric acid derivatives are metabolized in the liver via uridine 5'-diphosphate-glucuronosyl transferase enzymes (UGT), which are induced by the HIV PI ritonavir. Indeed, ritonavir significantly lowers plasma concentrations of other drugs metabolized by this enzymatic system by 40-50 percent. As UGT activity is induced, the metabolism of UGT substrates (gemfibrozil) will increase, resulting in a decrease in their plasma concentrations. Preliminary data in non-HIV-infected subjects suggest that reduced plasma concentrations of gemfibrozil are likely to result in reduced efficacy of the drug. Despite the fact that many HIV-infected patients with hypertriglyceridemia are likely to be receiving triglyceride-lowering therapy with a fibric acid derivative while simultaneously receiving antiretroviral therapy that includes ritonavir (i.e. lopinavir + ritonavir [LPV/r]), these two drugs have not been studied in combination to determine whether or not they interact. The objective of this study is to characterize the impact of LPV/r on the pharmacokinetic (PK) profile of gemfibrozil, after a single 600 mg oral dose, administered to healthy volunteers. In a longitudinal study design, fifteen subjects will receive a single, 600 mg dose of gemfibrozil before and after 13 days of LPV/r 400/100 mg twice daily. Gemfibrozil pharmacokinetics will be determined on days one and 14 and compared using the student t-test. Results from this study will provide (or refute) the rationale for further studies designed to assess the possibility of dose-adjusting gemfibrozil when it is given in combination with ritonavir in order to maximize the pharmacologic effects of gemfibrozil.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age of 18 to 65 years.
* Healthy by medical history and physical exam.
* Test HIV negative.
* Screening laboratory values within institutional normal range.
* Negative serum pregnancy test for females of child-bearing potential within 7 days prior to the initiation of LPV/r.
* Willingness and ability of females of child-bearing potential to practice abstinence or use effective non-hormonal methods of birth control (i.e. condom, diaphragm, IUD, spermicide, etc.) during the study.
* Non-smoker for at least 6 weeks prior to study participation. Subjects who are not currently smoking must refrain from smoking during the entire study period.

EXCLUSION CRITERIA:

* Concomitant routine therapy with any prescription, over-the-counter, herbal, or holistic medications, including oral contraceptives for 30 days prior to study participation.
* Subjects taking oral contraceptives currently, or within 30 days prior to study initiation.
* Intermittent (PRN) use of acetaminophen, non-steroidal antiinflammatory medications (i.e. ibuprofen), and loperamide will be allowed during the study.
* Subjects will be allowed to take a multivitamin with minerals, or equivalent, once daily if they desire to do so.
* Inability to obtain venous access for sample collection.
* Known presence of diabetes mellitus, human immunodeficiency virus (HIV) infection, active tuberculosis, cardiac disease (hypertension; congestive heart failure etc.), renal disease (chronic or acute renal failure or insufficiency), thyroid disease, hepatitis, respiratory disease (uncontrolled asthma or chronic obstructive pulmonary disease), myasthenia gravis, glaucoma, or uncontrolled peptic ulcer disease. Any other condition that may interfere with the interpretation of the study results or that may not be in the best interest of the subject in the opinion of the investigator.
* Positive pregnancy test or breastfeeding female.
* The presence of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
* Drug or alcohol use that may impair safety or adherence.
* History of intolerance or allergic reaction (rash; hives; swollen lips; difficulty breathing) to fibric acid derivatives (e.g. gemfibrozil, fenofibrate, bezafibrate, etc.) or protease inhibitors (ritonavir, lopinavir; indinavir, nelfinavir, saquinavir, atazanavir, fosamprenavir, darunavir, tipranavir).
* Inability or unwillingness of females of child-bearing potential to use a non-hormonal (barrier) method of contraception throughout the study (e.g. condom; diaphragm, etc.).
* Non-fasting total cholesterol or triglycerides greater than or equal to 270 mg/dL.
* Participation in another study during the entire study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Penzak, Pharm.D., Principal Investigator — CC Pharmacy Department
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Result] Busse KH, Hadigan C, Chairez C, Alfaro RM, Formentini E, Kovacs JA, Penzak SR. Gemfibrozil concentrations are significantly decreased in the presence of lopinavir-ritonavir. J Acquir Immune Defic Syndr. 2009 Oct 1;52(2):235-9. doi: 10.1097/QAI.0b013e3181b0610e. PMID 19648824

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Up to 30 healthy volunteers will be screened to enroll a total of 15 healthy volunteers. We will actively encourage participation of all ethnic groups and females. Recruitment of HIV-negative volunteers will be done through the normal volunteer office at NIH.
Pre-assignment Details: Subjects who meet inclusion criteria and do not meet any exclusion criteria will be invited to participate in the study.
Groups:
- Gemfibrozil (GF) Alone Followed by GF+ Lopinavir-ritonavir: Subjects received a single 600 mg dose of gemfibrozil before and after receiving lopinavir-ritonar 400mg/100mg twice daily, for 14.5 days. After each gemfibrozil dose, blood samples were collected to determine gemfibrozil plasma concentrations. These plasma concentrations were then used to determine gemfibrozil pharmacokinetic (PK) parameter values such as area under the concentration vs. time curve (AUC). Gemfibrozil PK parameter values were then compared before- and after lopinavir-ritonavir administration.
Period: Overall Study
Arm/Group | Gemfibrozil (GF) Alone Followed by GF+ Lopinavir-ritonavir
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Gemfibrozil (GF) Alone Followed by GF + Lopinavir-ritonavir: Subjects received a single 600 mg dose of gemfibrozil before- and after receiving lopinavir-ritonar 400mg/100mg twice daily, for 14.5 days. After each gemfibrozil dose, blood samples were collected for the determination of gemfibrozil plasma concentrations. The plasma concentrations were then used to determine gemfibrozil pharmacokinetic (PK) parameters values such as area under the concentration vs. time curve (AUC). PK Parameter values were then compared pre- and post lopinavir-ritonavir administration.
Arm/Group | Gemfibrozil (GF) Alone Followed by GF + Lopinavir-ritonavir
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Gemfibrozil Area Under the Concentration vs. Time Curve (AUC)
Description: AUC (ng*hr/mL) of gemfibrozil when given as a 600 mg dose by itself compared to gemfibrozil AUC after 14.5 days of lopinavir-ritonavir (400mg/100mg) twice daily.
Time Frame: 22 days per subject (approximately 1 year for entire study completion)
Population: Fifteen healthy volunteers were enrolled in this protocol based on an a priori power analysis. All 15 subjects completed the protocol and results reported are those from all 15 participants.
Measure: Geometric Mean (90% Confidence Interval); unit: ng*hr/mL
Groups:
- Gemfibrozil Alone (Control Group): Subjects received a single 600 mg dose of gemfibrozil and serial blood samples were collected over a 24 hr. post-dose period to determine pharmacokinetic parameter values. Area under the concentrations vs. time curve from time zero to infinity (i.e. total drug exposure) was the primary pharmacokinetic parameter of interest. After completing participation in this control group, each subject "crossed over" to received lopinavir-ritonavir (400mg/100mg twice daily) for 14.5 days. Therefore, each subject served as their own control. Hence there were two groups of data analyzed, but each group consisted of the same subjects (tested under different conditions).
- Gemfibrozil + Lopinavir-ritonavir: After receiving lopinavir-ritonavir (400mg/100mg twice daily) for 14.5 days, subjects received a single 600 mg dose of gemfibrozil and serial blood samples were collected over a 24 hr. post-dose period to determine pharmacokinetic parameter values. Area under the concentrations vs. time curve from time zero to infinity (i.e. total drug exposure) was the primary pharmacokinetic parameter of interest.
Arm/Group | Gemfibrozil Alone (Control Group) | Gemfibrozil + Lopinavir-ritonavir
Number analyzed (Participants) | 15 | 15
ng*hr/mL | 104 [90 to 118] | 62 [55 to 68]
Statistical Analysis 1: Comparison: Gemfibrozil Alone (Control Group) vs Gemfibrozil + Lopinavir-ritonavir; Null hypothesis: lopinavir-ritonavir does not alter gemfibrozil pharmacokinetics. A sample size of 13 healthy subjects yielded 81% power to detect a clinically relevant change of 30% in gemfibrozil AUC with concomitant lopinavir-ritonavir (alpha = 0.05; beta = 0.2). Gemfibrozil pharmacokinetic parameters derived pre- and post lopinavir-ritonavir exposure (Days 1 and 14, respectively) were compared using a paired Students t test; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Students paired, two-tailed T-test

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study. Each subject particpiated in this study for approximately 22 days, while the entire duration of the study (collectively) for all 15 subjects was approximately one year.
Arm/Group | Gemfibrozil (GF) Alone Followed by GF + Lopinavir-ritonavir
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes